CLINICAL TRIAL: NCT04718571
Title: Nontuberculous Mycobacteria Identified in Clinical Samples in the Geneva Area Over a Period 2015-2020
Brief Title: An Ecological Analysis of Nontuberculous Mycobacteria in the Geneva Area (2015-2020)
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Professor Jean-Paul Janssens, University Hospital, Geneva
Other Study IDs: 2020-00872
Record Dates: First submitted 2020-12-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Ecology of Nontubercuous Mycobacteria; Geneva Area

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of NTM diseases has been increasing regularly over the past 30 years in industrialized countries Although NTM are identified worldwide, there are important geographical disparities as to the relative prevalence of NTM species There are no data covering the ecology of NTM in Switzerland. Because of the progressive increase in NTM clinical cases in area Geneva(as noted in other industrialized countries), reporting the specific NTM distribution is important and relevant. In this study, the investigators aimed to: 1/ describe the relative prevalence of NTM species in clinical samples analyzed in the Geneva area, covering ca 500'000 inhabitants over a 5-year period; 2/ determine how many culture positive patients were treated; and 3/ specify the clinical sites involved.

DETAILED DESCRIPTION:
This study was performed in the Geneva University Hospitals (HUG), a 2008-bed complex providing care for a population of ca. 500'000 inhabitants. All clinical samples sent for microbiological analysis within HUG are treated by the Bacteriology Laboratory of Geneva University Hospitals. An online database is kept up-to-date and includes all samples processed by the laboratory. The investigators performed a comprehensive analysis of all clinical samples included in this database over a 5-year period (2015-2020). This report focuses only on positive results for nontuberculous mycobacteria (NTM).The following items were recorded: age, gender, BMI whenever available, site of infection (when pulmonary: description of main radiological abnormalities), presence and type of immunosuppression, relevant pulmonary and non-pulmonary comorbidities, results of microscopy, and NTM species identified. The investigators also recorded whether the patient was treated for the identified NTM or not and if a susceptibility profile had been determined (this is not routinely performed and must be requested by the clinician).

The study protocol was approved by their local ethics committee

ELIGIBILITY:
Inclusion criteria - patients with positive clinical samples for nontuberculous mycobacteria (NTM)

Exclusion criteria

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with positive clinical samples for nontuberculous mycobacteria (NTM)
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Identify nontuberculous mycobacteria species | 2015-2020
  Results of microscopy (positive or negative smear examination), and NTM species were identified (Rapidly or slow growing mycobacteria)

SECONDARY OUTCOMES:
Baseline characteristics of patients | 2015-2020
  Age (in years),
Baseline characteristics of patients | 2015-2020
  gender
Baseline characteristics of patients | 2015-2020
  BMI (in kg/m2)
Baseline characteristics of patients | 2015-2020
  site of infection (pulmonary or extrapulmonary)
Baseline characteristics of patients | 2015-2020
  presence and type of immunosuppression( HIV co-infection, chemotherapy, glucocorticoids)

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No